CLINICAL TRIAL: NCT04921462
Title: Silastic Sheet Usefulness Following Septoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Responsible Party: Principal Investigator, Leen Hijazi, Medical intern, King Abdulaziz Medical City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC20/509
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Septoplasty
Keywords: Intranasal splint; Silastic sheet; quilting suture; NOSE score

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silastic group (Active Comparator): included patients who underwent nasal septoplasty followed by insertion of silastic intranasal splint
  Interventions: Procedure: Septoplasty surgery
- Quilting group (Active Comparator): included patients who underwent septoplasty followed by quilting suture (Septal through and through suture)
  Interventions: Procedure: Septoplasty surgery

INTERVENTIONS:
Procedure: Septoplasty surgery — septoplasty procedures were performed by a single surgeon using the same technique among all patients. The procedures were conducted under general anesthesia according to the standard preoperative care used in our institution.

SUMMARY:
This study aimed to evaluate the effectiveness of silastic septal splint in reducing the rates of complications, decreasing the post-operative pain, and improving satisfaction in comparison to quilting suturing technique.

Methods:

A single center randomized controlled trial, including adult above the age of 18. A total of 50 participants who underwent septoplasty were enrolled and randomly assigned into two groups, Silastic group (n=25), and quilting group (n=25). Nasal obstruction severity was assessed by using an Arabic validated version of NOSE score, preoperatively then 3 days, one week and one month postoperatively. Post-operative complications were assessed at outpatient clinic 1 week and 1 month postoperatively. Pain was assessed by a 10-point numerical scales via phone call on the 3rd day postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) healthy individuals of both genders with deviated nasal septum and no other concomitant procedures.

Exclusion Criteria:

* 1. Concomitant procedure other than septoplasty. 2. Previous history of septal or nasal surgery. 3. Presence of nasal polyps, chronic sinusitis or other regional pathology. 4. Bleeding disorders or anticoagulation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Change in NOSE score 1 month postoperatively | 1 month postoperatively
  NOSE change = preoperative NOSE - 1 month postoperative NOSE

SECONDARY OUTCOMES:
Validated NOSE score | NOSE score preoperatively, 3 days, 1 week and 1 month postoperatively
complications | 1 month
  Bleeding, Bad smell, Synechia, Crustation and Perforation
postoperative pain | at 3 days postoperative
  using numerical Pain scale (0 to 10)
general satisfaction questionnaire | at 1 month postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical City, Riyadh, Saudi Arabia